CLINICAL TRIAL: NCT04422665
Title: Exercise 'Prehabilitation': A Novel Intervention to Protect Against Disuse-induced Muscle Atrophy and Sarcopenia in the Old
Brief Title: Preventing Bed-rest Induced Muscle Loss in the Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Birmingham (Other)
Collaborators: Biotechnology and Biological Sciences Research Council (Other); University of Nottingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: RG_16-100
Record Dates: First submitted 2020-06-01; First posted 2020-06-09 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-01

CONDITIONS: Muscle Loss; Disuse Atrophy; Protein Metabolism; Prehabilitation; Sarcopenia
MeSH Terms: conditions — Muscular Atrophy; Muscular Disorders, Atrophic; Sarcopenia | interventions — Resistance Training

STUDY DESIGN:
Intervention Model Description: Participants will be randomly allocated to one of two intervention groups. Due to the single-legged typed of resistance exercise, each subject will be its own control.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single Exercise (Experimental): Subjects allocated to this group will perform a single bout of one-legged resistance exercise. This bout will take place 1 day prior to the start of the bed rest. The resistance exercise will consist of 8 sets of leg extensions and 8 sets of leg curls. The non-exercising leg will serve as an internal control. The dominant leg will perform the exercise.
  Interventions: Other: Resistance exercise
- Multi Exercise (Experimental): Subjects allocated to this group will perform 4 bouts of one-legged resistance exercise. These bouts will take place on alternate days the week leading up to the bed rest. Each resistance exercise bout will consist of 8 sets of leg extensions and 8 sets of leg curls. The non-exercising leg will serve as an internal control. The dominant leg will perform the exercise.
  Interventions: Other: Resistance exercise

INTERVENTIONS:
Other: Resistance exercise — Single-legged resistance exercise

SUMMARY:
Episodes of inactivity due to hospitalisation, as short as 5 days, are associated with rapid muscle and strength loss in the elderly. The observed muscle loss with inactivity is likely due to muscle anabolic resistance and increased breakdown rates of muscle tissue. This is of great concern as the average hospital stay in the elderly is 5-6 days. Moreover, minor illnesses not requiring hospitalisation generally require short-term periods of inactive home-based recovery. The accumulation of repeated disuse events in older individuals manifests in a chronic muscle anabolic resistance (i.e. the inability of muscle to respond to anabolic stimuli such as exercise and nutrition) that may underpin the slow but devastating process of age-related muscle loss.

It is our belief that strategies to promote muscle health in ageing and reduce healthcare expenditure, should focus on alleviating muscle deterioration and anabolic resistance during short-term disuse.

In this regard, we propose that resistance exercise (i.e. weight lifting) performed prior to a disuse event (termed 'prehabilitation') may be sufficient to offset muscle loss in older individuals. Thus, we suggest the potent effect of resistance exercise in older muscles may prevent muscle loss during short-term disuse.

DETAILED DESCRIPTION:
Participants will be assigned to either single-bout (SINGLE; n=10) or multiple-bouts (MULTI; n=10) of resistance exercise prehabilitation prior to 5 consecutive days of bed rest. Groups will be matched for age, anthropometric characteristics and activity levels. Only males will be studied due to potential gender differences in muscle protein turnover. A single-leg resistance exercise prehabilitation model will allow for a direct within-subject comparison against the non-exercised control leg.

Preliminary Assessments

Following an induction meeting and obtainment of informed consent, participants will report to The National Institute of Health/Wellcome Trust Clinical Research Facility (CRF) at University Hospital Birmingham (UHB) at 0800h having fasted from 2100h the previous night. After measuring height and weight, the following parameters will be determined in the order outlined:

1. Muscle biopsy, blood and saliva sampling: a muscle biopsy sample will be obtained from a specific thigh muscle under local anaesthetic. A blood sample will then be obtained from a forearm vein. Participants will also provide a saliva sample. This will be obtained prior to the following measurements.
2. Lower-limb function: The short physical performance battery (SPPB) test will be used.
3. Body composition: bioelectrical impedance analysis will be used to determine fat/fat-free mass on a whole-body and anatomical regional basis (CRF nurse).
4. Muscle size/architecture: The thickness of the thigh muscles will be determined via non-invasive ultrasound imaging.
5. Leg strength and muscle activation: Estimated maximal leg strength will be measured firstly on a standard knee extension exercise machine.
6. Stable isotope procedure: Immediately following muscle biopsy, blood and saliva sampling, participants will orally consume a small bolus of 'heavy water' tracer to label the body water pool with a small amount of this isotope. Participants will provide a daily saliva sample to monitor body water tracer enrichment. This technique will allow us to quantify muscle protein synthesis over the course of prehabilitation and bed-rest.
7. Participants will be fitted with an accelerometer and pedometer to asses daily activity levels.
8. Participants are given a food diary to record daily nutritional intake over a 3-day period.

Exercise Prehabilitation (Days 0-7) Participants will be randomly assigned to undergo 4 resistance exercise bouts the week before (Day 1, 2, 5 and 7), or 1 resistance exercise bout on the evening prior to bed rest (i.e. Day 7). Exercise bouts will consist of 8 sets of single-leg knee extension exercise and 8 sets of single-leg leg curls. The non-exercised control leg will remain passive throughout training. Resistance exercise will be performed at 70% of previously determined maximal strength (10-15 repetitions).

Intervention - 5-days of bed-rest (Days 8-13) Participants will report to the CRF at 0700h the morning immediately after exercise prehabilitation phase. At 0800h, muscle biopsies will be obtained from both legs to assess changes in muscle metabolism over the 7 days of prehabilitation. Participants will then be transported for dual energy x-ray absorptiometry (DXA), Magnetic Resonance Imaging (MRI) and ultrasound assessment of body/muscle composition, after which the 5 consecutive days of strict bed rest will begin. The bed rest model will mimic a traditional inpatient hospital stay and reflect the level of muscle unloading that occurs in older individuals following acute illness. Participants will spend the majority of time in bed and will be allowed to adjust the hospital bed head height for reading, eating and watching television, but will otherwise be instructed to lie flat in bed. Bathing/hygiene will be performed in a wheelchair at a sink. The bathroom accessed using a wheelchair. Adherence to bed rest will be monitored by nursing staff and through daily analysis of accelerometry data.

Post Intervention Assessments (Day 13) On the morning after completion of the 5-day bed rest phase (i.e. Day 13) participants will awake at 0700h in the CRF and remain in bed for assessment of muscle protein synthesis in trained and untrained control legs. A cannula will be inserted into a vein of both forearms for frequent blood sampling and a stable isotope tracer infusion. During the tracer infusion, muscle biopsies will be obtained from both trained and untrained legs before and after consumption of a milk protein drink, to assess muscle metabolism. Participants will then be transported by wheelchair for repeat bioelectrical impedance analysis, MRI and ultrasound scans to assess body/muscle composition. Leg strength will be reassessed in trained and untrained legs. A physiotherapist will perform a functional assessment of participants before they are discharged.

Rehabilitation Training Participants will be given the opportunity to complete a 6-week rehabilitation programme, consisting of a progressive 3 x weekly leg resistance training with protein supplementation, designed to fully restore any loss in muscle mass and strength from short-term bed rest. Resistance training rehabilitation will not form a specific study objective, but muscle size and strength will be assessed to ensure restoration of any muscle decline from bed rest.

ELIGIBILITY:
Inclusion Criteria:

* Males aged between 65-80 years
* No history of structured resistance training within 10 years prior to study participation.
* Generally good health as indicated by a thorough health questionnaire.
* A score of ≥9 points on the Short Physical Performance Battery to assess lower extremity function.
* Body Mass Index <30kg/m2

Exclusion Criteria:

* Coagulation disorders
* Myocardial infarction
* Artery/vein disease
* Hormone replacement therapy
* Other chronic/systemic illnesses (i.e. renal failure, chronic obstructive pulmonary disease, cancer).
* Undergone 2 or more muscle biopsies from each leg previously.
* Received a stable isotope infusion in the last 3 years prior to study enrollment.

Ages: 65 Years to 80 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
Integrated myofibrillar protein synthesis rates | 2 years
  Myofibrillar protein synthesis rates will be measured during the prehabilitation and bed rest period in both the exercising and resting leg.
Muscle mass via MRI | 2 years
  Muscle volume in the quadriceps will be assessed before and after bed rest using magnetic resonance imaging techniques

SECONDARY OUTCOMES:
Muscle fibre properties | 2 years
  Via immunohistochemical staining procedures muscle fibre cross sectional area will be determined
Physical activity levels | 2 years
  Daily average time spent in sedentary, light, moderate or vigorous intensity activity using an accelerometer
Step-count | 2 years
  activity will be determined using accelerometry. Furthermore, step count will be Daily step-count assessed using a hip-worn pedometer
Plasma biomarkers of metabolic health | 2 years
  Blood markers - serum total cholesterol, serum high-density lipoprotein cholesterol, serum non-high-density lipoprotein cholesterol, total cholesterol, serum non-esterified fatty acids, serum triglycerides (units of measure for all - mmol/L)
Serum insulin | 2 years
  Via ELISA kits, resting insulin will be assessed using baseline plasma samples from before and after the bed rest period (pmol/l)
Intramuscular signaling via western blot | 2 years
  Western blots for phosphorylation of key anabolic and catabolic signaling proteins will be performed.
Gene expression | 2 years
  Search Results Web results
  Reverse transcription polymerase chain reaction (RT-PCR) will be performed to assess gene-expression of muscle anabolic and catabolic genes.
Dietary intake | 2 years
  Dietary intake will be assessed using 3-day weighed food diaries.
Body composition | 2 years
  Bioelectrical impedance analysis will be used to determine whole body fat and fat-free mass (units are % of total body mass for both fat and fat-free mass).
Leg strength | 2 years
  Estimated maximal leg strength will be determined for the leg extension and leg curl before and after the bed rest period
Height | 2 years
  measured using a stadiometer (cm)
Body weight | 2 years
  Measured using a digital weighing scale (kg)
Body Mass Index | 2 years
  Weight and height will be combined to report BMI in kg/m^2

CONTACTS AND LOCATIONS:
Locations (1):
- University of Birmingham, School of Sport, Exercise and Rehabilitation Sciences, Edgbaston, West Midlands, United Kingdom

IPD SHARING:
Plan to Share IPD: No